CLINICAL TRIAL: NCT05026619
Title: Youth Outlook on Life Opportunities Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Poh Lin Tan, Assistant Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: NUS-IRB-2020-362
Record Dates: First submitted 2021-08-16; First posted 2021-08-30 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Childbearing, Delayed; Marriage Age; Educational Problems; Anxiety; Age Related Female Infertility
MeSH Terms: conditions — Reproductive Behavior; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Placebo Comparator): Receives a fact sheet on diabetes in Singapore
  Interventions: Other: Information about diabetes
- Fertility-related information (Experimental): Receives accurate information on age-related fertility
  Interventions: Other: Information about age-related fertility
- Policy-related information (Experimental): Receives accurate information on local policy initiatives related to age at marriage and childbearing
  Interventions: Other: Information about policy initiatives

INTERVENTIONS:
Other: Information about age-related fertility — The following information is provided:
  Age and fertility IVF success rates and side effects
  Arms: Fertility-related information
Other: Information about policy initiatives — The following information is provided:
  Assisted reproductive technology treatment subsidies Other fertility-related policies
  Arms: Policy-related information
Other: Information about diabetes — The following information is provided:
  Diabetes risk factors and treatment Diabetes-related policies
  Arms: Control

SUMMARY:
Singapore's fertility rate is currently below 1.2, raising concerns about population ageing and long-term sustainability. The fertility decline is characterized by falling birth rates among women in their 20s with almost no recuperation among women in their 30s. This project explores a) whether informational imperfections help to account for high intended ages at childbearing in Singapore, b) whether informational interventions significantly affect ideal and expected ages at marriage and childbearing, and expected probability of undergoing social egg freezing, and c) whether informational interventions significantly affect expected and actual educational outcomes and labor market outcomes.

Our hypotheses are:

1. University students have knowledge gaps about age-related onset of infertility, assisted reproductive technologies and local policy initiatives related to age at marriage and childbearing, especially among male students.
2. Being exposed to accurate information in these domains leads to significantly lower ideal/expected ages at marriage and childbearing, and higher expected probability of undergoing social egg freezing, immediately after the intervention.
3. Being exposed to accurate information in these domains does not lead to lower educational and labor market expectations immediately after the intervention among either male or female students, or to significant differences in module choices, Cumulative Average Point (CAP), starting salary and employment status of university students in the following academic semester and six months after graduation, among either male or female students.

DETAILED DESCRIPTION:
The project conducts a randomized controlled trial involving 1000 full-time undergraduate students at NUS. The trial has three stages.

In the first stage, participants will be recruited through campus advertisements.

In the second stage, participants who meet the eligibility criteria will complete a 30-40 minute online survey. The survey includes the following:

1. a background survey on items including age, race, family income and parental background,
2. a section on dating history,
3. questions on ideal/expected ages at marriage, expected probability of undergoing social egg freezing, and fertility and educational and career expectations,
4. a section on mental wellbeing,
5. an awareness survey on age-related onset of infertility, assisted reproductive technologies, and local policy initiatives related to age at marriage and childbearing,
6. an informational intervention. One-third of participants (333 individuals) are randomly assigned to receive accurate information on the age-related fertility survey items. One-third of participants (333 individuals) are randomly assigned to receive accurate information on policy-related survey items. One-third of participants (334 individuals) receives a fact sheet on diabetes in Singapore. Participants are asked to read the information thoroughly,
7. selected questions from c), which collects data on after-intervention intended ages at marriage and fertility and educational and career expectations, as well as questions about whether the questions were useful or led to anxiety.

In the third stage, the students' responses are linked to the Educational Data Lake managed by ALSET, Provost's Office, NUS, which collects data on students' module choices (whether within the same major, in a different major within the same faculty or in a different faculty) and CAP in the following academic semester and at graduation, graduation status, and starting salary and employment status six months after graduation. All participants are informed and these linkages are mentioned in the consent form.

After the data collection is completed, we will analyse the data using a difference-in-differences econometric model. Our model compares three sets of dependent variables at different points in time:

1. Ideal/expected ages at marriage and fertility, expected probability of undergoing social egg freezing, and educational and career expectations, compared before and immediately after the intervention,
2. Module choices and CAP, compared before the survey and in the following academic semester and at graduation, and graduation status,
3. Starting salary and employment status, compared between the control and treatment groups six months after graduation (multiple regression rather than difference-in-differences model)

The results are compared by gender, faculty, educational and career expectations, and other background characteristics, including dating history and mental wellbeing.

ELIGIBILITY:
Inclusion Criteria:

* Full-time NUS undergraduate
* Singaporean citizen
* Aged 20-24
* Never been married
* Childless and not currently expecting
* Identify as heterosexual

Exclusion Criteria:

- Student enrolled in faculty where the Dean has not provided approval for recruitment

Ages: 20 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1000 (Actual)
Dates: Start 2021-09-21 (Actual); Primary Completion 2021-10-02 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Ideal age at marriage (both self and future spouse), first birth and number of children | Within one year and two years of initial survey
  During initial survey: Continuous
Expected age at marriage (both self and future spouse), first birth and number of children | Within one year and two years of initial survey
  During initial survey: Continuous percent chance by the following ages A. 25 B. 30 C. 35 D. 40
Expected probability of undergoing social egg freezing (only for females respondents) | Within one year and two years of initial survey
  During initial survey: Continuous percent chance of social egg freezing if available at the following ages:
  A. 25 B. 30 C. 35 D. 40

SECONDARY OUTCOMES:
Expected levels of education (both self and future spouse) | Within one year and two years of initial survey
  During initial survey: Continuous percent chance:
  A. Less than Bachelor's Degree B. Bachelor's Degree or higher C. Master's Degree or higher D. Doctoral Degree or higher
Expected earnings (both self and future spouse) | Within one year and two years of initial survey
  During initial survey: Continuous at the following ages:
  A. 25 B. 30 C. 35 D. 40
Expected full-time working status | Within one year and two years of initial survey
  During initial survey: Continuous percent chance by the following ages A. 25 B. 30 C. 35 D. 40
Expected occupation (self) at age 35 | Within one year and two years of initial survey
  During initial survey: Continuous percent chance:
  A. Full-time homemaker B. Manager or administrator in a private company C. Manager or administrator in the government/education sector D. Professional without doctoral degree (e.g. engineer, architect, accountant, social worker, teacher) E. Professional with doctoral degree or equivalent (lawyer, physician, scientist, college professor) F. Sales (e.g. insurance agent, real estate) G. Other (e.g. small business owner, etc.)
Expected contribution to housework and childcare if married with young children | Within one year and two years of initial survey
  During initial survey: Continuous percentage
Usefulness and anxiety over information presented | Within one year and two years of initial survey
  During initial survey: Strongly disagree, Disagree, Neither agree nor disagree, Agree, Strongly agree
Cumulative Point Average (CAP) | Within two years and six years of initial survey
  Measured in the following academic semester and at graduation
Module choices | Within two years and six years of initial survey
  Whether within the same major, in a different major within the same faculty or in a different faculty, in the following academic semester and at graduation
Graduation and honours | Within six years of initial survey
  Whether graduated and class of honours
Employment status six months after graduation | Within six years of initial survey
  Whether employed, full-time status
Starting salary | Within six years of initial survey
  Continuous

CONTACTS AND LOCATIONS:
Overall Officials: Poh Lin Tan, PhD, Principal Investigator — National University of Singapore
Locations (1):
- National University of Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
The collected data, data catalogue and research materials (i.e. study protocol, informed consent form, survey items) will be made available to researchers at the National University of Singapore (NUS) through the ALSET Data Lake within five years of the conclusion of the research project. Data will remain available for at least 10 years after any publication making use of the data. The ALSET Data Lake is managed by the NUS Instituted for Applied Learning Sciences and Educational Technology and operated by NUS IT. Questions about accessing the data from parties outside NUS can be sent to the PI or alsdl@nus.edu.sg.
Supporting Information: Study Protocol, ICF
Time Frame: The research data will be made available through the ALSET Data Lake within five years of the conclusion of the research project. Data will remain available for at least 10 years after any publication that makes use of the data.
Access Criteria: Approval from ALSET, Provost's Office, NUS-IRB and in compliance with Singapore's Personal Data Protection Act